CLINICAL TRIAL: NCT03181906
Title: Effectiveness of Pre-Consultation Medication Reconciliation Service in Reducing Unintentional Medication Discrepancies During Transition of Care From Hospital Discharge to Primary Care Setting- A Randomised Controlled Trial
Brief Title: Effectiveness of Pre-Consultation Medication Reconciliation Service in Reducing Unintentional Medication Discrepancies During Transition of Care From Hospital Discharge to Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Kee Kok Wai, Dr., National Healthcare Group, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DSRB2015/01219
Record Dates: First submitted 2017-06-02; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Medication Administered in Error; Medication Adherence
Keywords: medication discrepancy; primary care; transition of care
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Consultation Medication Reconciliation (Experimental): Participants underwent medication reconciliation service before their consultation with the attending doctor. A best possible medication history (BPMH) was created and saved as an electronic draft in the electronic medical record system.
  Interventions: Other: Pre-Consultation Medication Reconciliation
- Control (No Intervention): Participants in the control group proceeded with usual care, where the doctor reviewed the patient's condition and ordered an electronic prescription

INTERVENTIONS:
Other: Pre-Consultation Medication Reconciliation — Medication reconciliation service to be done for participants randomised to the intervention group
  Arms: Pre-Consultation Medication Reconciliation

SUMMARY:
This study evaluates the the effectiveness of pre-consultation Medication Reconciliation Service in reducing unintentional medication discrepancies among patients who discharged from hospital to primary care.

DETAILED DESCRIPTION:
Medication discrepancies during care transition were common. Many factors contribute to the risk of medication discrepancies. Despite medication reconciliation service being practiced in the hospital setting, there was limited knowledge on its effectiveness in the primary care setting. This study aims to evaluate the effectiveness of a pre-consultation medication reconciliation service in reducing medication discrepancies in patients who transit from hospital to primary care. Adult patients who made their first visit to the polyclinics following a recent hospital discharge and were prescribed with 5 or more chronic medications were randomised to 2 groups. Pre-consultation medication reconciliation by a pharmacist was carried out for the intervention group. Outcome was assessed by a different pharmacist who was blinded to the randomised allocation. The control group underwent usual care without a pre-consultation medication reconciliation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years and older
2. Patient or primary caregiver was able to provide informed consent
3. Patient or primary caregiver was English, Mandarin or Malay speaking
4. Patient was able to self-administer medications, or accompanied by a caregiver who assisted in administering medications
5. Patient was prescribed 5 or more chronic medications
6. The day of the study visit was the first follow-up visit in National Healthcare Group Polyclinics for chronic disease management after recent discharge from a local public hospital

Exclusion Criteria:

1. Residents of nursing home
2. The day of the study visit was for acute illness consult
3. Unwilling to consent to a 30-day follow-up phone call.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Unintentional medication discrepancies | 1 day
  Any unintentional medication discrepancies after doctor's consultation

SECONDARY OUTCOMES:
Types of medication discrepancies | 1 day
  Type of medication discrepancies, by a validated instrument by Claeys et al, (Claeys C, Neve J, Tulkens PM, Spinewine A. Content Validity and Inter-Rater Reliability of an Instrument to Characterize Unintentional Medication Discrepancies.Drugs & Aging. 2012 July; 29(7): 577-91.)
Causes of medication discrepancies | 1 day
  Causes of medication discrepancies, by a validated instrument by Claeys et al, (Claeys C, Neve J, Tulkens PM, Spinewine A. Content Validity and Inter-Rater Reliability of an Instrument to Characterize Unintentional Medication Discrepancies.Drugs & Aging. 2012 July; 29(7): 577-91.)
Medication adherence | 30 days
  Medication adherence by The 8-item Morisky Medication Adherence Scale
30-day re-hospitalisation | 30 days
  rate of re-hospitalisation 30 days after the study visit

CONTACTS AND LOCATIONS:
Overall Officials: Kok Wai Kee, MMED, Principal Investigator — National Healthcare Group Polyclinics

IPD SHARING:
Plan to Share IPD: Undecided